CLINICAL TRIAL: NCT05400330
Title: Long-Term Follow-Up to Evaluate the Safety of LX1001 in Participants With APOE4 Homozygote Alzheimer's Disease
Brief Title: Long-Term Follow-up of Gene Therapy for APOE4 Homozygote Alzheimer's Disease
Acronym: LEADLTFU
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Lexeo Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LX1001-02
Record Dates: First submitted 2022-05-27; First posted 2022-06-01 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Previously administered LX1001 (Experimental): This is a long-term follow-up study to evaluate the safety following LX1001, a gene therapy, for participants who are APOE4 homozygotes with clinical diagnoses varying from MCI or dementia due to AD who have previously received LX1001. Study LX1001-01 was designed to assess the safety of LX1001 at 4 ascending doses (1.4 × 1010, 4.4 × 1010, 1.4 × 1011 gene copy [gc]/mL CSF and 1.4 x 1014 [fixed dose]) as per droplet digital polymerase chain reaction methodology, with each group consisting of approximately n=3-5 individuals for a total of approximately 15 participants for the entire study.
  In this study, participants who have received LX1001 in the parent protocol (LX1001-01) will be followed for up to 260 weeks post gene therapy administration
  Interventions: Biological: LX1001

INTERVENTIONS:
Biological: LX1001 — Gene therapy
  Other Names: AAVrh.10hAPOE2

SUMMARY:
The primary purpose of this long-term follow-up study is to assess the long-term safety profile of APOE4 homozygote participants who were administered gene therapy (LX1001) for the treatment of Alzheimer's disease in Study LX100101. A secondary objective is to assess the biomarker as shown by the conversion of CSF APOE isoforms from APOE4 to APOE2-APOE4. Additional secondary outcomes include amyloid PET scan, CSF markers (including Aβ42, Aβ42/Aβ40 ratio T--tau, and P-tau), and quantitative MRI (and other biomarkers that may be informative for this therapeutic approach). Other secondary objectives include instruments to assess cognitive and clinical AD and to evaluate if treatment with AAVrh.10hAPOE2 improves brain tau pathology with tau PET scan (LX1001-01 Cohorts 3 and 4 only).

DETAILED DESCRIPTION:
This is a long-term follow-up study to evaluate the safety following LX1001, a gene therapy, for participants who are APOE4 homozygotes with clinical diagnoses varying from MCI or dementia due to AD who have previously received LX1001. Study LX1001-01 was designed to assess the safety of LX1001 at 4 ascending doses (1.4 × 1010, 4.4 × 1010, 1.4 × 1011 gene copy [gc]/mL CSF and 1.4 x 1014 [fixed dose]) as per droplet digital polymerase chain reaction methodology, with each group consisting of approximately n=3-5 individuals for a total of approximately 15 participants for the entire study.

In this study, participants who have received LX1001 in the parent protocol (LX1001-01) will be followed for up to 260 weeks post gene therapy administration to assess the safety and efficacy parameters (~208 weeks within this study)

ELIGIBILITY:
Inclusion Criteria:

* Participants who received LX1001 in study LX1001-01

Exclusion Criteria:

* Participants with any clinically significant medical condition that, in the opinion of the investigator, would pose a risk to participant safety
* Participants who agree not to post their personal medical data in relation to this study or any study information online, including social media sites, until all participants have completed all LX1001 clinical studies, including long-term follow-up.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-05-08 (Actual); Primary Completion 2028-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment emergent adverse events | 260 weeks
  All emergent adverse events will be collected
Incidence of serious adverse events | 260 weeks
  All incidents of serious adverse events will be collected

CONTACTS AND LOCATIONS:
Overall Officials: Lexeo Clinical Trials, Study Director — Lexeo Therapeutics
Locations (2):
- United States (2):
  - PPD- Orlando Research Unit, Orlando, Florida
  - Duke University, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: No